CLINICAL TRIAL: NCT04442971
Title: Investigation of the Effectiveness of Music Therapy on the Level of Consciousness of Neurological Early Rehabilitation Patients
Brief Title: Effectiveness of Music Therapy on Level of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOC-MT
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neurologic Disorder; Traumatic Brain Injury; Disorder of Consciousness
Keywords: neurological rehabilitation; music therapy; level of consciousness; default mode network
MeSH Terms: conditions — Nervous System Diseases; Brain Injuries, Traumatic; Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Music Stimulation (Experimental): Patients preferred music is presented via headphones.
  Interventions: Behavioral: Music Stimulation
- Alternative Auditory Stimulation (Active Comparator): An audio book is presented via headphones.
  Interventions: Behavioral: Alternative Stimulation
- No Auditory Stimulation (Sham Comparator): Silence is presented via headphones.
  Interventions: Behavioral: No Auditory Stimulation

INTERVENTIONS:
Behavioral: Music Stimulation — Patients wear headphones for 30 minutes/day over a period of four weeks and listen to their preferred music.
  Arms: Music Stimulation
Behavioral: Alternative Stimulation — Patients wear headphones for 30 minutes/day over a period of four weeks and listen to an audio book.
  Arms: Alternative Auditory Stimulation
Behavioral: No Auditory Stimulation — Patients wear headphones for 30 minutes/day over a period of four weeks and hear silence.
  Arms: No Auditory Stimulation

SUMMARY:
It is known that even in patients with severe disorders of consciousness (DOC), the perception of known stimuli triggers emotional reactions that can be interpreted as an expression of a residual function of consciousness. Music therapy has a long tradition in neurological rehabilitation. Frequently, active therapies with own music making and singing are implemented in clinical settings. In DOC patients, it is more likely to use passive music listening. However, findings on effectiveness are limited, as only a few studies have systematically investigated the effects of music therapy in this population. Therefore, the investigators want to investigate the effectiveness of passive listening to preferred music on the level of consciousness.

DETAILED DESCRIPTION:
Due to continuous improvements in acute medical care, the number of patients surviving severe brain damage has increased over the past decades. While some patients improve significantly during the first days after the injury, other patients remain in altered states of consciousness (i.e. coma, unresponsive wakefulness syndrome or minimally conscious state). In patients with disorders of consciousness (DOC), the auditory modality is preferably examined because the responsiveness within the motor and visual modality is often difficult to assess or impaired. Music is a special type of auditory stimulation that can be of particular benefit in DOC patients. The positive effects of music are attributed to the restoration of specific brain networks that are necessary for processing sensory inputs, as well as the emotional aspects of music, which can increase arousal and activate the reward system. Previous studies have shown that music, including passive listening to music, is associated with psychological and physical changes in both healthy and clinical populations. For example, listening to preferred music can reduce pain and anxiety and the need for sedation in different patient groups.

Music therapy has a long tradition in neurological rehabilitation. In DOC patients, passive listening to music is used (in contrast to active therapies used in fully conscious patients). Efficacy results are inconsistent, however, since only a few studies have systematically investigated the effects of music therapy. In previous investigations, either the sample size is very small or no control conditions have been used. A study that met both quality criteria was published by Sun & Chen in 2015. The authors compared two groups: while the music group (n = 20) listened to their favorite music for 15 to 30 minutes three times a day for a period of four weeks, the control group received no stimulation. Although the GCS values increased significantly in both groups, the music group showed a significantly stronger improvement in the level of consciousness. Based on this study, the present study wants to compare the effectiveness of passive listening to music with two control conditions (alternative auditory stimulation and no auditory stimulation) in early neurological rehabilitation patients.

It is a prospective, double-blind, controlled and randomized intervention study that is carried out monocentrically. Over a period of 24 months, 66 patients undergoing early neurological and neurosurgical rehabilitation after severe brain damage are included. For the individual patient, the study duration is a maximum of 38 days (preliminary phase: 3-7 days; intervention phase: 28 days; follow-up phase: 1-3 days). Patients are randomly assigned to one of three study arms (1. Musical stimulation; 2. Alternative auditory stimulation, 3. No auditory stimulation). In the preliminary phase (days 1 to 7), a native MRI (without contrast agent) and a CRS-R assessment are performed. In addition, there is a neurophysiological examination in which evoked potentials are recorded. In the subsequent main phase, the intervention takes place: Over a period of 28 days, the study participants wear headphones for 30 minutes a day, through which they are presented with preferred music (experimental arm), an audio book (comparative arm) or silence (control arm). In the main phase, a CRS-R test is carried out weekly to record the current state of consciousness. In the follow-up phase (1 to 3 days), the (native) MRI examination, the CRS-R assessment and the neurophysiological examination are repeated. The primary outcome measure is an improvement of the level of consciousness, measured with the Coma-Recovery-Scale-Revised (CRS-R).

ELIGIBILITY:
Inclusion Criteria:

* early neurological rehabilitation (phase B)
* traumatic brain injury
* disorder of consciousness (coma, UWS, MCS)
* at minimum two weeks after disease onset
* admission to intensive care unit
* written consent from the patient's legal representative
* Exclusion of pregnancy

Exclusion Criteria:

* insufficient cardiorespiratory stability
* fractures or severe infratentorial brain injuries leading to impaired auditory evoked potentials
* previous brain damage
* Known mental disorders (dementia, depression)
* hearing loss or deafness in one or two ears
* wounds that do not allow you to wear headphones
* colonization with multi-resistant pathogens
* MRI contraindications
* claustrophobia
* weight>120 kg

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in level of consciousness | 4 weeks
  Level of consciousness is measured with the Coma-Recovery-Scale-Revised (Range: 0 to 23) before and after treatment.

SECONDARY OUTCOMES:
Change in connectivity within the default mode network | 4 weeks
  Patients undergo a MRI scan before and after intervention. Each MRI scan has a duration of 30 minutes. Functional and structural sequences are measured. The resting-state scan (important for the assessment of the default mode network) has a duration of eight minutes and is performed without external stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, MD, Study Director — BDH-Clinic Hessisch Oldendorf; Melanie Boltzmann, PhD, Principal Investigator — BDH-Clinic Hessisch Oldendorf
Locations (1):
- BDH-Clinic Hessisch Oldendorf, Hessisch Oldendorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Period of availability begins when results are published, at the earliest in Dec 2022
Access Criteria: IPD can be obtained from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Kotchoubey B, Pavlov YG, Kleber B. Music in Research and Rehabilitation of Disorders of Consciousness: Psychological and Neurophysiological Foundations. Front Psychol. 2015 Nov 27;6:1763. doi: 10.3389/fpsyg.2015.01763. eCollection 2015. PMID 26640445
- [Background] Perrin F, Castro M, Tillmann B, Luaute J. Promoting the use of personally relevant stimuli for investigating patients with disorders of consciousness. Front Psychol. 2015 Jul 30;6:1102. doi: 10.3389/fpsyg.2015.01102. eCollection 2015. PMID 26284020
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Background] Sun J, Chen W. Music therapy for coma patients: preliminary results. Eur Rev Med Pharmacol Sci. 2015 Apr;19(7):1209-18. PMID 25912580